CLINICAL TRIAL: NCT07257874
Title: Comparison Between Intra-Operative Pectoral Block and Intravenous Analgesia for Post-Operative Pain Relief in Patients Undergoing Modified Radical Mastectomy
Brief Title: Intraoperative Pectoral Block vs IV Analgesia for Pain After Modified Radical Mastectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: No.179/IMDC/IREB-2025
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Mastectomy, Modified Radical
MeSH Terms: interventions — Bupivacaine; Injections; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECs Arm (Experimental)
  Interventions: Drug: bupivacaine 0.5% injection
- IV Analgesia Arm (Active Comparator)
  Interventions: Drug: Ketorolac 30 mg IV

INTERVENTIONS:
Drug: bupivacaine 0.5% injection — Intra-Operative Pectoral Block in Patients Undergoing Modified Radical Mastectomy for Post operative Pain management
  Arms: PECs Arm
Drug: Ketorolac 30 mg IV — Ketorolac 30mg administered Intravenously as a standard practice for post operative pain management in modified radical mastectomy
  Arms: IV Analgesia Arm

SUMMARY:
There is difference in post operative pain between patients receiving inter- pectoral block and those receiving standard Intravenous analgesia(INJ TORADOL) in patients undergoing Modified Radical Mastectomy.

To compare between these two methods , which one is better for post operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients undergoing Modified Radical Mastectomy for biopsy proven Carcinoma Breast
* Patient with age 18-65 years
* Patients with ASA Grade 2
* BMI less than 40 kg/meter square

Exclusion Criteria:

* Block site infection
* Coagulopathies (INR > 1.6 and Platelets < 100000)
* Any Organ dysfunction such as severe cardiac, pulmonary, renal or liver dysfunction
* Systemic infection
* Dementia
* Known hypersensitivity to local anesthetic agents

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Severity at 24 hours Measured by Numeric Pain Rating Scale from 0-10 , where 0 is no pain and 10 is severe pain. | 24 hours Post Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Akbar Niazi Teaching Hospital, Islamabad, Pakistan